CLINICAL TRIAL: NCT03583853
Title: Autophagy Genes and Interleukin-10 in Systemic Lupus Erythematosus Patients
Brief Title: Autophagy in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Mostafa, principle investigator, Assiut University
Other Study IDs: amkmm
Record Dates: First submitted 2018-06-22; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: take 5 ml blood for isolation of peripheral blood mono-nuclear cells then extraction of Ribonucleic acid (RNA) to determine the expression of autophagy genes by real time polymerase chain reaction (real time PCR)
  Interventions: Device: real time PCR
- control: take 5 ml blood for isolation of peripheral blood mono-nuclear cells then extraction of RNA to determine the expression of autophagy genes real time polymerase chain reaction
  Interventions: Device: real time PCR

INTERVENTIONS:
Device: real time PCR — real time PCR will be used for determination of expression of autophagy genes

SUMMARY:
Systemic lupus erythematosus is systemic autoimmune disease characterized by a wide range of clinical manifestations, from skin and mucosal lesions to severe injuries in the central nervous system, kidneys and other organs. The presence of high titres of autoantibodies against nuclear components, immune complexes deposition, complement deficiency and lymphocytes infiltration in affected tissues, which causes tissue and organ damage are the main characteristics of the disease. Nowadays, many studies elucidate the essential role of autophagy in the occurrence, development and severity of systemic lupus erythematosus.

DETAILED DESCRIPTION:
Autophagy is a highly conserved lysosome-mediated catabolic process. It can remove unwanted cytoplasmic components, such as long-lived and/or misfolded proteins, damaged organelles, playing an important role in maintaining cellular homeostasis and cell survival in stress conditions, such as nutrient deprivation and hypoxia.

Recently, Autophagy is implicated in nearly all steps of both innate and adaptive immune responses, including neutrophil extracellular trap and inflammasome formation, pathogen recognition, lymphocyte and monocyte development and function, antigen processing and presentation, type I interferon production and inflammatory regulation, thus playing an important part in maintaining the balance of immune system.

Autophagy is divided into three major types: macroautophagy, microautophagy, and chaperone-mediated autophagy, with macroautophagy being the most investigated and understood. Disturbances in autophagy have been implicated in chronic inflammatory diseases and several autoimmune diseases, including Systemic lupus erythematosus, multiple sclerosis, Crohn's disease and rheumatoid arthritis.

Several regulatory factors that may play key roles in autophagy processes have been discovered in recent years, such as beclin1, which is the key regulatory factor in the autophagy startup process, microtubule-associated protein-light chain 3, autophagy-related gene 5, which are components of autophagosomes.

ELIGIBILITY:
Inclusion Criteria:

* patients who fulfilled at least four criteria of systemic lupus erythematosus according to American College of Rheumatology

Exclusion Criteria:

* Pregnancy or lactation.
* coexistence of other autoimmune diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SLE patients are evaluated according to the SLE disease activity index 2000 (SLEDAI) and classified into two groups, one having active disease and the other group with inactive disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the expression of autophagy genes in systemic lupus erythematosus patients group and control group | Baseline and 6 months
  the expression of autophagy genes will be measured by real time polymerase chain reaction

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ciccacci C, Perricone C, Alessandri C, Latini A, Politi C, Delunardo F, Pierdominici M, Conti F, Novelli G, Ortona E, Borgiani P. Evaluation of ATG5 polymorphisms in Italian patients with systemic lupus erythematosus: contribution to disease susceptibility and clinical phenotypes. Lupus. 2018 Aug;27(9):1464-1469. doi: 10.1177/0961203318776108. Epub 2018 May 14. PMID 29759048
- [Background] Klionsky DJ. Autophagy: from phenomenology to molecular understanding in less than a decade. Nat Rev Mol Cell Biol. 2007 Nov;8(11):931-7. doi: 10.1038/nrm2245. PMID 17712358
- [Background] Zhang Y, Morgan MJ, Chen K, Choksi S, Liu ZG. Induction of autophagy is essential for monocyte-macrophage differentiation. Blood. 2012 Mar 22;119(12):2895-905. doi: 10.1182/blood-2011-08-372383. Epub 2012 Jan 5. PMID 22223827
- [Background] Dang J, Li J, Xin Q, Shan S, Bian X, Yuan Q, Liu N, Ma X, Li Y, Liu Q. Gene-gene interaction of ATG5, ATG7, BLK and BANK1 in systemic lupus erythematosus. Int J Rheum Dis. 2016 Dec;19(12):1284-1293. doi: 10.1111/1756-185X.12768. Epub 2015 Sep 30. PMID 26420661
- [Background] Zhu L, Wang H, Wu Y, He Z, Qin Y, Shen Q. The Autophagy Level Is Increased in the Synovial Tissues of Patients with Active Rheumatoid Arthritis and Is Correlated with Disease Severity. Mediators Inflamm. 2017;2017:7623145. doi: 10.1155/2017/7623145. Epub 2017 Feb 1. PMID 28255205
- [Background] Teruel M, Alarcon-Riquelme ME. The genetic basis of systemic lupus erythematosus: What are the risk factors and what have we learned. J Autoimmun. 2016 Nov;74:161-175. doi: 10.1016/j.jaut.2016.08.001. Epub 2016 Aug 10. PMID 27522116
- [Background] Zhou XJ, Lu XL, Lv JC, Yang HZ, Qin LX, Zhao MH, Su Y, Li ZG, Zhang H. Genetic association of PRDM1-ATG5 intergenic region and autophagy with systemic lupus erythematosus in a Chinese population. Ann Rheum Dis. 2011 Jul;70(7):1330-7. doi: 10.1136/ard.2010.140111. PMID 21622776
- [Background] Godsell J, Rudloff I, Kandane-Rathnayake R, Hoi A, Nold MF, Morand EF, Harris J. Clinical associations of IL-10 and IL-37 in systemic lupus erythematosus. Sci Rep. 2016 Oct 6;6:34604. doi: 10.1038/srep34604. PMID 27708376
- [Background] Lopez P, Alonso-Perez E, Rodriguez-Carrio J, Suarez A. Influence of Atg5 mutation in SLE depends on functional IL-10 genotype. PLoS One. 2013 Oct 18;8(10):e78756. doi: 10.1371/journal.pone.0078756. eCollection 2013. PMID 24205307
- [Background] Ward MM, Marx AS, Barry NN. Comparison of the validity and sensitivity to change of 5 activity indices in systemic lupus erythematosus. J Rheumatol. 2000 Mar;27(3):664-70. PMID 10743805